CLINICAL TRIAL: NCT03833544
Title: Effect of Lower Limb Flexor Synergy Training on Motor Function in Chronic Stroke - An Exploratory Study
Brief Title: Lower Limb Flexor Synergy Training in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist Rehabilitation Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRC_StrFlxTraining
Record Dates: First submitted 2019-02-04; First posted 2019-02-07 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2023-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Exercise training: Progressive resistance training of hip, knee, and ankle flexors.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Progressive resistance training of hip, knee, and ankle flexors.

SUMMARY:
This study evaluates whether a 4-week exercise training program focusing on lower limb flexors can improve lower limb motor function late after stroke. It is hypothesized that there would be significant improvements in gait and strength of the flexor muscles as a result of the training. It is also hypothesized that the training effects, if any, would be retained at 4 weeks after ending the training.

DETAILED DESCRIPTION:
It is known that the muscles that flex the hip, knee, and ankle joints are responsible for bringing the leg up and forward during walking and for a successful recovery from a slip or trip. Many previous studies have focused on strengthening the lower limb muscles that support the body in standing and walking (the so-called anti-gravity extensor muscles) but the training targeting the lower limb flexors has rarely been emphasized in stroke rehabilitation. Therefore, it is the intent of this exploratory study to find out whether an exercise training program focusing on lower limb flexors can improve lower limb motor function late after stroke.

Ten participants with chronic stroke will be recruited. Their lower limb muscle function and walking performance will be assessed at baseline (2 to 3 times within the 2 weeks prior to starting the training), at the end of training, and 4 weeks later.

Each subject will perform biking exercises under supervision, 2-3 times per week for 4 weeks (30 minutes each). The bike pedals are moving backward at a preset speed regardless of user effort. With feet strapped to the pedals, the participant will be asked to activate the hip, knee, and ankle flexors simultaneously when the pedal is moving up and then relax. Heart rate (HR) will be monitored continuously using a fingertip pulse monitor to ensure the maximum training HR is no more than 75% of the subject's HR Reserve.

ELIGIBILITY:
Inclusion Criteria:

* Time post-stroke between 6 months and 3 years
* Able to walk with or without an assistive device for 7 m independently
* Abnormal flexor synergy in both hip and knee joints (score 1 or 2) on the Fugl-Meyer Assessment Lower Extremity section II: Volitional movement within synergies (Fugl-Meyer et al., 1975)
* Walk slower than 1 m/s
* Able to understand and follow simple instructions
* Agree not to participate in strength training or supervised physical therapy during and for at least 4 weeks after the completion of training
* Previous participation in the physical therapy program for stroke without experiencing excessive symptoms (shortness of breath, headache, prolonged fatigue)

Exclusion Criteria:

* Current symptomatic coronary artery disease or congestive heart failure
* History of myocardial infarction
* Uncontrolled hypertension (>150/90 mm Hg)
* Lower limb fracture in the past 6 months
* Lower limb joint or muscular problems
* Acute or terminal illness
* Current participation in strength training or supervised physical therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Changes in Speed During Overground Gait | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  To test if the training can improve gait speed during overground walking, gait speeds will be obtained using a video-based 3D motion capture system before and after the training. To test if the gait speed changes are maintained after training, a follow-up test will be performed 4 weeks after training finished.
Changes in Speed During Obstacle Crossing | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  To test if the training can improve the speed during obstacle crossing (stepping over a 4x1.5x60 cm^3 wooden block), speeds during obstacle crossing will be obtained using a video-based 3D motion capture system before and after the training. To test if the speed changes are maintained after training, a follow-up test will be performed 4 weeks after training finished.
Changes in Step Length During Overground Gait | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  To test if the training can improve the step length during overground walking, step lengths will be obtained using a video-based 3D motion capture system before and after the training. To test if the step length changes are maintained after training, a follow-up test will be performed 4 weeks after training finished.
Changes in Step Length During Obstacle Crossing | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  To test if training can improve the step length during obstacle crossing (stepping over a 4x1.5x60 cm^3 wooden block), step lengths during obstacle crossing will be obtained using a video-based 3D motion capture system before and after the training. To test if the step length changes are maintained after training, a follow-up test will be performed 4 weeks after training finished.
Changes in Toe Clearance During Overground Gait | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  To test if the training can improve toe clearance during overground walking, toe clearances will be obtained using a video-based 3D motion capture system before and after the training. To test if the toe clearance changes are maintained after training, a follow-up test will be performed 4 weeks after training finished.
Changes in Toe Clearance During Obstacle Crossing | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  To test if the training can improve the toe clearance during obstacle crossing (stepping over a 4x1.5x60 cm^3 wooden block), toe clearances during obstacle crossing will be obtained using a video-based 3D motion capture system before and after the training. To test if the toe clearance changes are maintained after training, a follow-up test will be performed 4 weeks after training finished.
Changes in Peak Knee Flexion Angle in the Swing Phase During Overground Gait | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  To test if training can improve the peak knee flexion angle in the swing phase during overground walking, knee flexion angles will be obtained using a video-based 3D motion capture system before and after the training. To test if the angle changes are maintained after training, a follow-up test will be performed 4 weeks after training finished.
Changes in Peak Knee Flexion Angle in the Swing Phase During Obstacle Crossing | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  To test if the training can improve the peak knee flexion angle in the swing phase during obstacle crossing (stepping over a 4x1.5x60 cm^3 wooden block), knee flexion angles will be obtained using a video-based 3D motion capture system before and after the training. To test if the angle changes are maintained after training, a follow-up test will be performed 4 weeks after training finished.

SECONDARY OUTCOMES:
Changes in Muscle Activation Profiles During Overground Gait | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  To test if training can alter the lower limb muscle activation profiles during overground walking, surface electromyographic (EMG) signals of different lower extremity muscles during walking will be obtained using a wireless EMG system before and after the training. To test if the changes in profile are maintained after training, a follow-up test will be performed 4 weeks after training finished.
Changes in Muscle Activation Profiles During Obstacle Crossing | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  To test if the training can alter the lower limb muscle activation profiles during obstacle crossing (stepping over a 4x1.5x60 cm^3 wooden block), surface electromyographic (EMG) signals of different lower extremity muscles during obstacle crossing will be obtained using a wireless EMG system before and after the training. To test if the changes in profile are maintained after training, a follow-up test will be performed 4 weeks after training finished.
Changes in 6-min Walk Distance | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  In a 6-min walk test, the participant will be asked to walk back and forth around 2 small cones that are 30-m apart as fast as possible for 6 minutes. To test if the training can improve the walk distance in 6 minutes, the distances will be assessed before and after the training. To test if the changes in walk distance are maintained after training, a follow-up test will be performed 4 weeks after training finished.
Changes in Muscle Strength | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  To test if the training can improve muscle strength, isometric strength will be assessed in the hip flexors, knee flexors, and ankle dorsiflexors, bilaterally, using a Biodex System 3 dynamometer before and after the training. To test if the changes in muscle strength are maintained after training, a follow-up test will be performed 4 weeks after training finished.
Changes in Force Steadiness | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  During a force steadiness test, the participant will be asked to produce a knee flexion torque In the seated position as steady as possible for 10 seconds and match the target torque (10%, 30%, or 50% of maximum torque) displayed on a video monitor. To test if the training can improve the ability to hold a steady force, the force steadiness will be assessed before and after the training. To test if the changes in force steadiness are maintained after training, a follow-up test will be performed 4 weeks after training finished.
Changes in Lower Extremity Motor Function | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  The lower extremity motor function section of the Fugl-Meyer Assessment (Fugl-Meyer et al., 1975) (FMA-LEM) has a maximum score of 34 points (the higher the score the better the function). To test if the training can improve lower extremity motor function, FMA-LEM scores will be assessed by a licensed therapist before and after the training. To test if the changes in score are maintained after training, a follow-up assessment will be performed 4 weeks after training finished.
Changes in Spasticity | Weeks 1-2: Baseline Assessment (2-3 times); Weeks 3-6: Training (no assessment); Week 7: Post-training Assessment (within 1 week after the end of training); Week 10: Follow-up Assessment (4 weeks after the end of training)
  The Modified Ashworth scale (MAS) measures resistance during passive soft-tissue stretching and is a reliable scale for the assessment of spasticity in clinical settings (Bohannon and Smith, 1987). The MAS score ranged from 0 (no increase in muscle tone) to 5 (rigid muscle). To test if the training can improve spasticity, MAS scores of bilateral hip flexors, knee flexors, and ankle dorsiflexors will be assessed by a licensed therapist before and after the training. To test if the changes in score are maintained after training, a follow-up assessment will be performed 4 weeks after training finished.

CONTACTS AND LOCATIONS:
Overall Officials: John W Chow, PhD, Principal Investigator — Methodist Rehabiliation Center
Locations (1):
- Methodist Rehabilitation Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616